CLINICAL TRIAL: NCT04995458
Title: Clinical Evaluation of Cerasmart Implant-supported Posterior Crowns
Brief Title: Clinical Evaluation of Composite-ceramic Implant-supported Posterior Crowns (Cerasmart)
Acronym: Cerasmart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: GC Europe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC Europe N.V-4156360
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Dental Materials
Keywords: implant-supported crowns; monolithic zirconia; composite-ceramic; clinical evaluation; survival

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Composite-ceramic (Experimental): To assess the clinical performance and survival of posterior composite-ceramic implant-supported crowns
  Interventions: Procedure: composite-ceramic
- Monolithic zirconia (Active Comparator): To assess the clinical performance and survival of posterior monolitihic zirconia implant-supported crowns
  Interventions: Procedure: Monolithic zirconia

INTERVENTIONS:
Procedure: composite-ceramic — To assess the clinical performance of composite-ceramic crowns
  Other Names: Cerasmart
  Arms: Composite-ceramic
Procedure: Monolithic zirconia — To assess the clinical performance of monolithic z¡irconia crowns
  Arms: Monolithic zirconia

SUMMARY:
The objectives of the present study are to analyze and to compare the survival rates and possible biological and technical complications arising from the use of composite-ceramic posterior implant-supported crowns with those obtained when using their counterparts prepared using monolithic zirconia restorations. The null hypothesis is that no differences would be found between the parameters studied for each type of restoration.

DETAILED DESCRIPTION:
Eighty patients in need of posterior implant-supported crowns (n=80) were recruited from the Master of Buccofacial Prostheses and Occlusion, Faculty of Odontology, University Complutense of Madrid, Madrid, Spain. Before treatment, all participants were informed of the purpose of the study, the clinical procedures, the material to be used, and the advantages and risks of the restorations. They were asked to give their written informed consent to participate in the study.

Eighty posterior implant-supported crowns were produced and allocated in parallel an randomly to either monolithic zirconia or composite-ceramic restorations by means of a randomization list. A total of 40 implant-supported crowns were placed using monolithic zirconia and 40 composite-ceramic. The clinical procedures were performed by two experienced clinicians. Full-arch impressions were taken using addition silicone. The restorations were cemented using a resin-based cement. The occlusion was adjusted and the surfaces polished after cementing. All restorations were prepared by an experienced technician. The restorations will be examined at one week (baseline), 1, 2, and 3 years by two researchers who were not involved in the restorative treatment. Each assessor evaluated the restoration independently, and the worst assessment will be used in the event of discrepancies.

ELIGIBILITY:
Inclusion Criteria:

* One posterior tooth (molar or premolar) to restore, and with opposing tooth

Exclusion Criteria:

* unacceptable oral hygiene
* bruxism

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Quality of restorations at baseline | Baseline
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 1 year | 1 year
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 2 year | 2 years
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Quality of restorations at 3 year | 3 years
  The quality of the surface and color, anatomical form and marginal integrity was assessed using the California Dental Association's (CDA) assessment system. Each CDA criterion was ranked on a scale of 1 to 4, where 4 = excellent, 3 = good, 2 = unacceptable (repair), and 1 = unacceptable (replacement).
Plaque Index (PI) at baseline | baseline
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 1 year | 1 year
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 2 years | 2 years
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Plaque Index (PI) at 3 years | 3 years
  Plaque Index (PI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at baseline | Baseline
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 1 year | 1 year
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 2 years | 2 years
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Gingival Index (GI) at 3 years | 3 years
  Gingival Index (GI) of the abutment and control teeth. A score of 0 to 3 was assigned. Higher score means a worse outcome.
Probing depth at baseline | Baseline
  Probing depth of the abutment. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 1 year | 1 year
  Probing depth of the abutment. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 2 year | 2 years
  Probing depth of the abutment. A score of 0 to 4 was assigned. Higher score means a worse outcome
Probing depth at 3 year | 3 years
  Probing depth of the abutment teeth. A score of 0 to 4 was assigned. Higher score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: MARIA J SUAREZ, PhD, Study Director — Universidad Complutense de Madrid
Locations (1):
- Faculty of Odontology, Madrid, Spain